CLINICAL TRIAL: NCT01983761
Title: A Phase I/IIa, Open-label, Non-randomized, Study of ASC-101 in Patients With Hematologic Malignancies or Myelodysplastic Syndrome (MDS) Who Are Candidates for Dual-cord Umbilical Cord Blood Transplantation (UCBT)
Brief Title: Study of ASC-101 in Patients With Hematologic Malignancies Who Receive Dual-cord Umbilical Cord Blood Transplantation
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Targazyme, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ASC-101-001
Record Dates: First submitted 2013-11-02; First posted 2013-11-14 (Estimated); Last update posted 2013-11-18 (Estimated); Status verified 2013-11

CONDITIONS: Blood And Marrow Transplantation; Leukemia; Lymphoma; Transplantation Infection; Myelodysplastic Syndrome (MDS); Non-Hodgkin's Lymphoma (NHL); Hodgkin's Lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma; Myelodysplastic Syndromes; Lymphoma, Non-Hodgkin; Hodgkin Disease | interventions — fludarabine; Clofarabine; Busulfan; Whole-Body Irradiation; Bone Marrow Purging; Mycophenolic Acid; Tacrolimus; Rituximab; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fludarabine, Clofarabine, Busulfan, ATG, TBI (Myeloablative) (Experimental): Fludarabine, Clofarabine, Busulfan, Anti-thymocyte Globulin (ATG), Total Body Irradiation (TBI) (Myeloablative) Day Treatment
  * Day0 Admit, IV hydration, rituximab 375 mg/m2 (B cell malignancy)
  * Day 1 Fludarabine 10 mg/m2, clofarabine 30 mg/m2, busulfan AUC 5,000
  * Day2 Fludarabine 10 mg/m2, clofarabine 30 mg/m2, busulfan AUC 5,000
  * Day3 Fludarabine 10 mg/m2, clofarabine 30 mg/m2, busulfan AUC 5,000
  * Day4 Fludarabine 10 mg/m2, clofarabine 30 mg/m2, busulfan AUC 5,000, rabbit ATG 1.25 mg/kg
  * Day5 Low-dose TBI 2 Gy in AM, rabbit ATG 1.75 mg/kg
  * Day6 Rest
  * Day7 Rest
  * Day8 Cord blood infusions
  Interventions: Drug: Fludarabine, Clofarabine, Busulfan, ATG, TBI (Myeloablative)
- Fludarabine, Melphalan, ATG (Reduced Intensity) (Experimental): Day Treatment
  * Day0 Admit, hydration
  * Day1 Fludarabine 40 mg/m2 IV
  * Day2 Fludarabine 40 mg/m2 IV, rabbit ATG 1.25 mg/kg
  * Day3 Fludarabine 40 mg/m2 IV, rabbit ATG 1.75 mg/kg
  * Day4 Fludarabine 40 mg/m2 IV and Melphalan 140 mg/m2 IV
  * Day5 Rest Day6 Cord blood infusions
  Interventions: Drug: Fludarabine, Melphalan, ATG (Reduced Intensity)

INTERVENTIONS:
Drug: Fludarabine, Clofarabine, Busulfan, ATG, TBI (Myeloablative)
  Other Names: Interventions:◦Drug: Fludarabine; ◦Drug: Mycophenolate mofetil; ◦Drug: Tacrolimus; ◦Procedure: Cord Blood Infusion; ◦Drug: Rituximab; ◦Drug: ATG; ◦Drug: Busulfan; ◦Drug: Clofarabine
  Arms: Fludarabine, Clofarabine, Busulfan, ATG, TBI (Myeloablative)
Drug: Fludarabine, Melphalan, ATG (Reduced Intensity)
  Other Names: Interventions:◦Drug: Melphalan; ◦Drug: Fludarabine; ◦Drug: Mycophenolate mofetil; ◦Drug: Tacrolimus; ◦Procedure: Cord Blood Infusion; ◦Drug: ATG
  Arms: Fludarabine, Melphalan, ATG (Reduced Intensity)

SUMMARY:
The goal of this clinical research study is to learn if it is safe and feasible to transplant patients with one of two units of cord blood that has been changed in the laboratory before it is given. Only patients with leukemia, lymphoma or myelodysplastic syndrome will be allowed on this study. The secondary goal is to obtain the preliminary efficacy outcome. Researchers also want to learn if using cord blood that has been changed can help to control the disease.

One cord blood unit will not be changed before it is administered to you. The cord blood unit that will be altered will be changed to use sugar that is found in small amounts in blood cells. It plays a role in telling transplanted cells where they should go in the body. Adding more sugars to the cord blood cells in the laboratory helps the cord blood cells find their way to the bone marrow faster. This process is called fucosylation.

"Conditioning" is the chemo and other medicines and will be given to patients to prepare to receive cord blood transplant cells. This prevents immune system from rejecting the cells. Conditioning will be started before the transplant.

ATG is a protein that removes immune cells that cause damage to the body.

Clofarabine is designed to interfere with the growth and development of cancer cells.

Fludarabine is designed to interfere with the DNA of cancer cells, which may cause the cancer cells to die. This chemotherapy is also designed to block your body's ability to reject the donor's bone marrow cells.

Melphalan and busulfan are designed to bind to the DNA of cells, which may cause cancer cells to die.

MMF and tacrolimus are designed to block the donor cells from growing and spreading in a way that could cause graft versus host disease (GVHD -- a condition in which transplanted tissue attacks the recipient's body). This may help to prevent GVHD.

Rituximab is designed to attach to cancer cells, which may cause them to die.

A Phase I study for treatment of patients (N=25) with hematologic malignancies and MDS who are candidates for dual-cord UCBT is ongoing at M.D. Anderson Cancer Center under an Investigator-initiated IND Application, E.J. Shpall, MD, PI. Since August, 2012, Preliminary results indicate that ASC-101 UCBT is well-tolerated and no ASC-101 related untoward adverse events have been observed. To date, the median time to neutrophil engraftment (N=9) is 15 days, and the median time to platelet engraftment (N=9) is 33 days. The trial remains ongoing.

DETAILED DESCRIPTION:
Central Venous Catheter Placement:

You will first have a central venous catheter (CVC) placed. A CVC is a sterile flexible tube that will be placed into a large vein while you are under local anesthesia. Your doctor will explain this procedure to you in more detail, and you will be required to sign a separate consent form for it.

The chemotherapy, some of the other drugs in this study, and the cord blood transplant will be given by vein through your CVC. Blood samples will also be drawn through your CVC. The CVC will remain in your body for about 2-5 months.

Study Plans:

If you agree to take part in this study, your doctor will choose one of the following 2 study plans based on the disease and your age and medical history.

Fludarabine/Clofarabine/Busulfan/Rituximab/Total Body Irradiation:

If you are between 1 and 80 years of age and can receive high-dose chemotherapy, and your doctor agrees, you will receive fludarabine, clofarabine, busulfan, ATG, total body irradiation, and possibly rituximab.

If you are receiving this study plan medication, blood may be drawn to check levels of busulfan 1 or more times over the 4-day course of treatment. No more than 1 teaspoon will be taken at each blood draw.

Day Treatment

* Day0 Admit, IV hydration, rituximab 375 mg/m2 (B cell malignancy)
* Day1 Fludarabine 10 mg/m2, clofarabine 30 mg/m2, busulfan AUC 5,000
* Day2 Fludarabine 10 mg/m2, clofarabine 30 mg/m2, busulfan AUC 5,000
* Day3 Fludarabine 10 mg/m2, clofarabine 30 mg/m2, busulfan AUC 5,000
* Day4 Fludarabine 10 mg/m2, clofarabine 30 mg/m2, busulfan AUC 5,000, rabbit ATG 1.25 mg/kg
* Day5 Low-dose TBI 2 Gy in AM, rabbit ATG 1.75 mg/kg
* Day6 Rest
* Day7 Rest
* Day8 Cord blood infusions

Fludarabine, Melphalan

Day Treatment

* Day0 Admit, hydration
* Day1 Fludarabine 40 mg/m2 IV
* Day2 Fludarabine 40 mg/m2 IV, rabbit ATG 1.25 mg/kg
* Day3 Fludarabine 40 mg/m2 IV, rabbit ATG 1.75 mg/kg
* Day4 Fludarabine 40 mg/m2 IV and Melphalan 140 mg/m2 IV
* Day5 Rest
* Day6 Cord blood infusions

Supportive Drugs:

Starting on Day -3, you will receive mycophenolate mofetil as a tablet by mouth 2 times a day. If you are not able to take the tablet by mouth, you will receive MMF by vein over 2 hours 2 times a day. If you do not have GVHD at Day 100 after your cord blood transplant, the dose of MMF will be gradually lowered. If you have GVHD, MMF may be stopped 7 days after the GVHD is controlled.

Starting on Day -2, you will receive tacrolimus by vein as a continuous (nonstop) infusion until you are able to take it by mouth. You will then take tacrolimus by mouth 2 times a day for about 6 months. After that, your tacrolimus dose may be gradually lowered if you do not have GVHD. Your doctor will discuss this with you.

Starting on Day 0, you will receive filgrastim (G-CSF) through a needle under the skin 1 time a day every day until your white blood count begins to recover. Filgrastim is designed to help cells in the bone marrow to divide, which helps raise white blood cells counts more quickly, lower fever, and decrease the risk of infection.

Study Visits:

At about 6 weeks, 3, 6, and 12 months after the transplant:

* You will have a physical exam.
* You will be checked for possible reactions to the transplant and study drugs, including GVHD.
* Blood (about 4 teaspoons) will be drawn for routine tests, to check for CMV antibodies, and for genetic tests to learn if the donor's cells have "taken". The routine blood tests will be repeated as often as the doctor thinks is needed.
* If the doctor thinks it is needed, you will have a bone marrow aspiration to check the status of the disease.

You will need to stay in the hospital for about 4 weeks. After you leave the hospital, you will continue as an outpatient in the hospital area, which means you will have to stay close enough to be able to come back for any visits for about 100 days after the transplant.

Length of Participation:

If the study suits you and you agree to join, you will be in it for one year after your transplant. You will be taken off study early if the disease gets worse, if intolerable side effects occur, if the cord blood is infected and cannot be transplanted, if you are unable to follow study directions, or if your doctor thinks it is in your best interest.

This is an investigational study. Fucosylation is not an FDA-approved process. It is currently being used for research purposes only. Fludarabine, busulfan, clofarabine, melphalan, mycophenolate mofetil, tacrolimus, and rituximab are FDA approved and commercially available to be given to patients with leukemia or lymphoma having a cord blood transplant. Total body irradiation is delivered using FDA-approved and commercially available methods.

Up to 25 patients will be enrolled in this study. All will be enrolled at M.D. Anderson Cancer Center, Scripps Green Hospital,University Hospitals Case Medical Center, and Texas Transplant Institute.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females: 1 to 80 years of age
2. Patients with AML, ALL, CML, CLL, MDS, NHL or HD:

   Patients with AML: first complete remission (CR1) with high-risk for relapse (e.g., high-risk cytogenetics, molecular mutation [FLT3, MEK, MLL, other] and/or persistent minimal residual disease by evidence of flow cytometry < 20% blasts in marrow), secondary leukemia from prior chemotherapy and/or arising from MDS, Langerhan's cell histiocytosis, second or third complete remission (CR2 or CR3) Patients with ALL: CR1 with Philadelphia chromosome or translocation 4;11, hypodiploidy, and/or persistent minimal residual disease by flow cytometry), secondary leukemia from prior chemotherapy, CR2 or CR3 Patients with CML: second chronic phase after failure or intolerant of tyrosine kinase inhibitors, or accelerated phase Patients with MDS: IPPS INT-1 or higher and failed prior therapy Patients with NHL: CR2 or CR3 following response to prior therapy, or relapse, including relapse following autologous HSCT Patients with HD: CR2 or CR3 following response to prior therapy, or relapse, including relapse following autologous HSCT
3. KPS of 80 or ECOG < 3 (age 12 years) or Lansky Play Performance Score of > 60% (age < 12 years). Eligibility for pediatric patients will be determined in conjunction with an Institutional pediatrician.
4. Laboratory data:

   ALT/AST < 2.0 times the upper limit of normal (ULN) Total bilirubin < 2.0 times ULN Creatinine < 1.6 mg/dL
5. Left ventricular ejection fraction (LVEF) ≥ 40%
6. Pulmonary function test (PFT) demonstrating diffusion capacity of lung for carbon monoxide (DLCO) ≥ 50% of predicted. For children < 7 years of age who are unable to perform PFT, oxygen saturation > 92% on room air by pulse oximetry allowed.
7. Patients must have 2 UCB unit available, each matched with the patient at 4, 5, or 6/6 collect all 10 HLA class I (serological) and II (molecular) antigens. Each UCB unit must contain a minimum dose of 1.5 x107 (red blood cell depleted) TNC per kg per cord pre-thaw. Information on HLA-C and DQ loci will be collected for future analysis.
8. Have a back-up cell source identified in case of engraftment failure. The source can be autologous, allogeneic (related or unrelated).
9. Negative beta HCG test in a woman with child bearing potential defined as not post-menopausal for 12 months or no previous surgical sterilization and willing to use an effective contraceptive measure while on study
10. Patient, or guardian, ability to provide written informed consent

Exclusion Criteria:

1. Prior allogeneic transplant
2. Patients with 6/6 HLA-matched sibling donors, 10/10 HLA-matched unrelated donors (MUD), or untimely availability of 10/10 HLA-MUD relative to need to take patient to transplant
3. Active, uncontrolled infection, decompensated congestive heart failure or pulmonary insufficiency requiring oxygen supplementation
4. Active central nervous system (CNS) disease in patients with a history of CNS malignancy
5. Any other medical intervention or other condition which, in the opinion of the Principal Investigator, could compromise adherence with study requirements
6. Known positive for human immunodeficiency virus (HIV), hepatitis B virus surface antigen (HBsAg), or hepatitis C virus (HCV) or rapid plasma regain (RPR) test for syphilis
7. Pregnant or breast-feeding
8. Treatment with any investigational product within 28 days prior to Screening

Ages: 1 Year to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2013-11; Primary Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability in patients who receive ASC-101-treated dual-cord UCBT | 42 days
  All safety endpoints will be summarized using descriptive statistics; no inferential testing is planned. For chimerism, graphic presentations of changes from baseline will be provided.

SECONDARY OUTCOMES:
Preliminary efficacy of ASC-101-treated dual-cord UCBT, as assessed by the rate of reconstitution of neutrophils and platelets as compared to historical controls receiving an unmanipulated dual-cord UCBT | 180 days
  The rate of reconstitution of neutrophils and platelets in the peripheral blood as compared to historical controls receiving an unmanipulated UCBT The rate and severity of aGVHD The rates of infectious complications and antibiotic usage The rate of disease relapse The rate of transplant-related mortality Days 100 and 180 disease-free and overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Shpall, MD, Study Chair — M.D. Anderson Cancer Center
Locations (4):
- United States (4):
  - Scripps Green Hospital, La Jolla, California
  - University Hospitals of Cleveland, Cleveland, Ohio
  - M.D. Anderson Cancer Center, Houston, Texas
  - Texas Transplant Institute, San Antonio, Texas